CLINICAL TRIAL: NCT04045080
Title: The Use of AMADEO in Hand Rehabilitation in Patients With Parkinson Disease
Brief Title: Hand Rehab Using AMADEO in PD Patients
Acronym: P-AMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Rocco Salvatore Calabrò, Medical Director, Neurologist, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 41/19
Record Dates: First submitted 2019-08-02; First posted 2019-08-05 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AMADEO Training (Experimental): Twenty PD patients with hand bradykinesia will be treated with the AMADEO® system. They will undergo 15 training sessions, 5 a week for 3 weeks, each session lasting about 60 minutes. During each session, both the hands will be treated using the endeffector in its active and active-assisted modality.
  Interventions: Device: AMADEO; Other: Training
- OT training (Active Comparator): Twenty control subjects (PD patients) will be treated with traditional rehabilitation focused on fine hand-finger movement skills. The patients in this group will undergo the same amount of treatment.
  Both the groups will be trained with conventional physiotherapy concerning postural, balance and gait.
  Interventions: Other: OT Training

INTERVENTIONS:
Device: AMADEO — AMADEO® is an end-effector system enables intensive training with frequently repeated gripping movements. It offers the possibility to select from between passive, assistive and active modes using exercise of finger strength, finger movement, movement control and a selective activation of the fingers.
  Moreover, even without muscular strength, active work can be done using EMG-based training. The Continuous Passive Motion (CPM Plus) therapy facilitates the implementation of automatic movement sequences even when the patient is unable to complete the entire range of motion on their own. It may be used in all phases of finger-hand rehabilitation and can be adapted to the needs of every patient.
  In patients with PD, it will be useful in improving bradykinesia and potentially distal hypostenia.
  Arms: AMADEO Training
Other: Training — training
  Arms: AMADEO Training
Other: OT Training — training
  Arms: OT training

SUMMARY:
Hand movements are particularly impaired in Parkinson's Disease (PD) patients contributing to functional disability and difficulties in activities of daily living. AMADEO®. is an end-effector system enables intensive training with frequently repeated gripping movements. It offers the possibility to select from between passive, assistive and active modes using exercise of finger strength, finger movement, movement control and a selective activation of the fingers.Aim of this study is to evaluate the efficacy of the end-effector finger system, AMADEO®, on hand-finger movements in PD patients evaluating the improvement on finger tapping and agility of hand movement item scores on the MDS-UPDRS, variation on the active finger strengths and the active and passive Range of Motion (ROM); variation on Electromyographic (EMG)-parameters.

ELIGIBILITY:
Inclusion Criteria

* Idiopathic PD diagnosed according to the Gelb's criteria;
* Hoehn-Yahr stage 1- 3
* "On" state
* MMSE score ≥ 24
* Willing and able to give written informed consent;
* Willing and able to comply with the study procedures.

Exclusion Criteria

* A specific kind of fluctuation: Sudden on-off fluctuations
* History sign or symptoms suggesting the diagnosis of atypical or secondary Parkinsonisms;
* History of stereotaxic brain surgery for PD;
* Mini-mental examination (MMSE) score less than 24 at screening;
* Changes in Levodopa (DA) dose in any time within 4 week prior to baseline;
* Changes in Dopamine Agonists (DA) in any formulation in any time within 4 week prior to baseline;
* Presence of severe dyskinesia prior to baseline;
* Any other medical or psychiatric condition that may compromise the patient's participation in this study;

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Nine hole peg test | 1 month
  9HPT is used to measure finger dexterity in patients with various neurological diagnoses

SECONDARY OUTCOMES:
Bipolar surface electromyography | 1 month
  EMG will be recorded from the first dorsal interossieous (FDI) and extensor digitorum communis (EDC) muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Rocco S Calabrò, Study Chair — IRCCS Centro Neurolesi
Locations (1):
- IRCCS Centro Neurolesi "Bonino-Pulejo", Messina, Italy

IPD SHARING:
Plan to Share IPD: No